CLINICAL TRIAL: NCT01554761
Title: Effect of Posterior Corneal Toricity on Refractive Outcome of Pseudophakia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Jinsong Zhang, MD,the President of Eye hosptial of China Medical Univerisity,China, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2012-02-27; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Astigmatism; Cataract
Keywords: astigmatism; pseudophakia
MeSH Terms: conditions — Astigmatism; Cataract; Pseudophakia | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: phacoemulsification — After topical anesthesia with Alcaine, 3.0-mm clear corneal incisions were made. Torsional phacoemulsification was performed using the Infiniti Vision System with the OZil handpiece, a 45-degree Kelman miniflared tip, and DuoVisc viscoelastic (all from Alcon).
Device: Pentacam (Oculus,Germany)examination — Total corneal astigmatism is obtained by Pentacam at every visit.

SUMMARY:
This study is to evaluate the necessity of considering posterior corneal toricity on refractive outcome of patients with cataracts and corneal astigmatism after implantation of intraocular lenses.

This is determined by comparing total corneal and refractive astigmatism,and by comparing the expected refractive result with actual refractive astigmatism postoperatively,using total corneal and anterior corneal astigmatism to calculate respectively.

ELIGIBILITY:
Inclusion Criteria:

* cataract candidates
* preoperative corneal regular astigmatism >0.75D
* Willing and able to complete all required postoperative visits
* Able to comprehend and sign a statement of informed consent

Exclusion Criteria:

* significant intraocular lenses tilt or decentration
* corneal scarring
* Irregular corneal astigmatism
* other ocular diseases
* surgical complication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Pentacam-derived corneal astigmatism | 3month postoperatively
refraction | 3month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Zhang, MD, Principal Investigator — Eye Hospital of China Medical University
Locations (1):
- Eye hospital of China Medical Univerisity, Shenyang, Liaoning, China